CLINICAL TRIAL: NCT00625326
Title: A Phase II Study of the Dose-Effect of COL-121 Ointment in Patients With Plaque-Type Psoriasis
Brief Title: Study of Dose-Effect of COL-121 Ointment in Patients With Plaque-Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deltanoid Pharmaceuticals (Industry)
Responsible Party: Michael Graeber, Head of Global Clinical Project Management & US Development, Galderma
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COL-121-PSOR-201
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Plaque-type Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 75 µg/g COL-121 Ointment (Experimental): 75 µg/g COL-121 Ointment
  Interventions: Drug: COL-121
- 150 µg/g COL-121 Ointment (Experimental): 150 µg/g COL-121 Ointment
  Interventions: Drug: COL-121
- 300 µg/g COL-121 Ointment (Experimental): 300 µg/g COL-121 Ointment
  Interventions: Drug: COL-121
- 50 µg/g Calcipotriene Ointment (Active Comparator): 50 µg/g Calcipotriene Ointment (active control)
  Interventions: Drug: 50 µg/g Calcipotriene Ointment
- Placebo Ointment (Placebo Comparator): Placebo Ointment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COL-121 — 75 µg/g COL-121 Ointment
  Arms: 75 µg/g COL-121 Ointment
Drug: 50 µg/g Calcipotriene Ointment — 50 µg/g Calcipotriene Ointment
  Other Names: Dovonex
  Arms: 50 µg/g Calcipotriene Ointment
Drug: Placebo — Placebo
  Arms: Placebo Ointment
Drug: COL-121 — 150 µg/g COL-121 Ointment
  Arms: 150 µg/g COL-121 Ointment
Drug: COL-121 — 300 µg/g COL-121 Ointment
  Arms: 300 µg/g COL-121 Ointment

SUMMARY:
Low doses of topically administered vitamin D analogs have been shown to have an anti-psoriatic effect without the risk of hypercalcemia. Calcipotriol, the most thoroughly studied of the vitamin D analogs, was first approved in Europe in the early 1990s. It has been shown to be comparable or slightly more effective than class II corticosteroid ointments. However, patients had reduced levels of parathyroid hormone; mean serum and urine calcium were increased during treatment and hypercalciuria was observed. These effects were reversible with discontinuation of therapy. Thus, while calcipotriol ointment was shown to be effective, the potential for alterations in calcium homeostasis have limited its use to 100 g of ointment per week (0.5 mg calcipotriol/week). Work has continued on the creation of new vitamin D analogs, such as COL-121, with the intent of eliminating the adverse effects of hypercalcemia and hypercalciuria with a compound that is more stable and more easily administered.

DETAILED DESCRIPTION:
Psoriasis affects more than 7 million Americans. Plaque-type psoriasis (the most common type of psoriasis) is an inflammatory skin condition with reactive abnormal epidermal differentiation and hyperproliferation. It is characterized by raised, thickened, plaques of erythematous skin covered by a silvery-white scale. Plaque-type psoriasis is most commonly found on the knees, elbows, and scalp but can appear anywhere on the body. While patients with psoriasis may complain of itchiness and discomfort, the psychological effects of the disease are the most debilitating. In a 1998 survey conducted by the National Psoriasis Foundation, it was found that 79% of the psoriasis patients surveyed reported that the disease had a negative impact on their lives and 40% felt frustrated with the ineffectiveness of their current therapies.

Although the exact cause of this skin disease is unknown, it is clear that immune-based inflammatory mechanisms initiate an accelerated growth of skin cells. This accelerated growth results in an agglomeration of skin cells on the surface of the epidermis that the body cannot shed. This agglomeration creates the thickened patches of scaly skin characteristic of the disease.

Clinical use of systemic vitamin D to treat psoriasis has been limited because of the induction of hypercalcemia. In contrast, low doses of topically administered vitamin D analogs have been shown to have an anti-psoriatic effect without the risk of hypercalcemia. Topical vitamin D analogs have the ability to inhibit the proliferation and promote the differentiation of keratinocytes in psoriatic skin. In addition, vitamin D analogs may also act by inhibiting cytokine production by keratinocytes or lymphocytes. Calcipotriol, the most thoroughly studied of the vitamin D analogs, was first approved in Europe in the early 1990s. It has been shown to be comparable or slightly more effective than class II corticosteroid ointments. In patients with extensive psoriasis, calcipotriol ointment was shown to be effective. However, patients had reduced levels of parathyroid hormone; mean serum and urine calcium were increased during treatment and hypercalciuria was recorded in 3 patients. These effects were reversible with discontinuation of therapy. In a review of the effects on calcium homeostasis, it was noted that calcipotriol (50 µg/g) had no effects on serum or urine calcium when administered at doses of 40-50 g/week and two reports of hypercalcemia at doses of 70-100 g/week. Thus, while calcipotriol ointment was shown to be effective, the potential for alterations in calcium homeostasis have limited its use to 100 g of ointment per week (0.5 mg calcipotriol/week). Subsequently, calcipotriol and tacalcitol, another vitamin D analog, have become first-line therapies in the management of "mild to moderate" psoriasis in several countries in Western Europe, Japan and the USA.

Work has continued on the creation of new vitamin D analogs, such as COL-121, with the intent of eliminating the adverse effects of hypercalcemia and hypercalciuria with a compound that is more stable and more easily administered.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis must affect at least 2% and not more than 10% of the subject's body surface area, excluding the face and scalp
* Subject must have 2 to 4 target plaques on the area to be treated, excluding the face and scalp.
* Subjects who are women of childbearing potential must have a negative pregnancy test and be non-lactating.
* Subjects who are women of childbearing potential must utilize one of the following methods of birth control throughout the study: IUD, diaphragm, a condom, a spermicidal gel or foam, oral contraceptives (provided subject has been utilizing this method for at least 4 months prior to Visit 1 and has not changed the brand within this period). Subjects may also participate if they are surgically sterilized, in a monogamous relationship with a sterile partner, or abstain from sexual intercourse during the course of the study.
* Subjects must be in good general health and free of any disease state or physical condition that, in the investigator's opinion, may interfere with study evaluations or exposes the subject to unacceptable risk by study participation.
* Subject must be willing and able to apply the study medication as directed, comply with the study instructions, and commit to all the follow-up visits for the duration of the study.
* Subjects must sign an informed consent form.

Exclusion Criteria:

* Subjects who have guttate, pustular, erythrodermic or other non-plaque types of psoriasis.
* Subjects who have spontaneously improving or rapidly deteriorating plaque psoriasis.
* Subjects who have used systemic immunomodulatory therapy known to affect psoriasis and to typically decrease immune cell populations (e.g., alefacept) within the previous 40 weeks.
* Subjects who have used any systemic immunomodulatory therapy known to affect psoriasis and to NOT typically decrease immune cell populations (e.g., etanercept) within the previous 16 weeks.
* Subjects who have used any photo-therapy (including laser), photo-chemotherapy or systemic psoriasis therapy (e.g., systemic corticosteroids, methotrexate, retinoids, cyclosporine) within the previous 12 weeks.
* Subjects who have had prolonged exposure to natural or artificial sources of ultraviolet radiation within the previous 3 weeks or are intending to have such exposure during the study, thought by the investigator likely to modify the subject's plaque psoriasis.
* Subjects who have used topical anti-psoriatic therapy (including topical retinoids) on the areas to be evaluated within the previous 2 weeks.
* Subjects who have used emollients/moisturizers on the areas to be evaluated within the previous 1 day.
* Subjects who have untreated bacterial, tubercular, fungal or viral lesions of the skin on the areas to be evaluated.
* Subjects who have known sensitivity to a component of the study medication or to topical or systemic vitamin D.
* Subjects who have any significant condition such as diseases of the hepatic, renal, endocrine, musculoskeletal, or nervous system, or any gross physical impairment.
* Subjects who have taken a vitamin D supplement that exceeds 400 IU per day in the previous 30 days.
* Subjects who have taken a calcium supplement that exceeds 1200 mg per day in the previous 30 days.
* Subjects who are using lithium or Plaquenil.
* Subjects who are using beta-blocking medication or thiazide diuretics whose dose has not been stable for at least 12 weeks.
* Subjects who have a history of hypercalcemia or evidence of vitamin D toxicity.
* Subjects who are currently being treated for malignancy or have been diagnosed with melanoma within the past 5 years.
* Subjects who have received any investigational treatment(s) within the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Physician's Global Assessment | Randomization and Day 84

SECONDARY OUTCOMES:
Change from Baseline of PGA score | Day 0, week 2, 4, 8, 12, and 16
  PGA score is a scale from 0 to 5, with 0=clear and 5=very severe
Change from baseline of Psoriasis Signs Severity (PSS) | Day 0, week 2, 4, 8, 12, and 16
  Psoriasis Signs Severity (PSS) is the investigator's evaluation of the severity of each of three key signs of psoriasis (erythema, plaque elevation, and scaling). The PSS for a target plaque is the sum of the individual sign scores for that target plaque. The Erythema Severity Scale, Plaque Elevation Severity Scale, and the Scaling Severity Score are each assessed on a scale from 0=clear to 5=very severe. These scores combined = PSS.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (20):
- United States (20):
  - East Bay Dermatology Medical Group, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Dermatology Specialists, Inc., Vista, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - The Savin Center, PC, New Haven, Connecticut
  - International Dermatology Research, Inc., Miami, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Dermatology Specialists, Louisville, Kentucky
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Northwest Cutaneous Research Specialists, Portland, Oregon
  - Philadelphia Institute of Dermatology, Flourtown, Pennsylvania
  - DermResearch, Inc., Austin, Texas
  - Dermatology Associates of San Antonio, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Premier Clinical Research, Spokane, Washington